CLINICAL TRIAL: NCT06493123
Title: "Postoperative Mobilization and Bottle-P.E.P. in Heart Valve Surgery:A Prospective Randomized Controlled Study "
Brief Title: Cardiopulmonary Rehabilitation In Heart Valve Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Dilek Unsal, Investigator, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Saglik Bilimleri University
Record Dates: First submitted 2024-05-08; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Heart Valve Diseases
Keywords: heart valve surgery; bottle-P.E.P.; early mobilization; cardiopulmonary rehabilitation
MeSH Terms: conditions — Heart Valve Diseases | interventions — Early Ambulation

STUDY DESIGN:
Intervention Model Description: * Group I/Control: Conventional cardiopulmonary rehabilitation will be applied in the postoperative period.
  * Group II/ Bottle P.E.P.: Conventional cardiopulmonary rehabilitation and bottle-PEP therapy will be applied in the postoperative period.
  * Group III/Early Mobilization: An early mobilization program will be started in conventional cardiopulmonary rehabilitation in the postoperative period.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Group I/Control group: Conventional cardiopulmonary rehabilitation will be applied in the postoperative period.
  Interventions: Other: Conventional Cardiopulmonary Rehabilitation
- Group II (Experimental): Group II/ Bottle P.E.P.: Conventional cardiopulmonary rehabilitation and bottle-PEP therapy will be applied in the postoperative period.
  Interventions: Other: Conventional Cardiopulmonary Rehabilitation; Other: Bottle P.E.P. (Pozitive Expiratory Pressure)
- Group III (Experimental): Group III/Early Mobilization: Early mobilization program will be started in conventional cardiopulmonary rehabilitation in the postoperative period.
  Interventions: Other: Conventional Cardiopulmonary Rehabilitation; Other: Early Mobilization

INTERVENTIONS:
Other: Conventional Cardiopulmonary Rehabilitation — Conventional cardiopulmonary applications including positioning, chest physiotherapy, in-bed normal joint movement exercises, sitting and walking, posture exercises
Other: Bottle P.E.P. (Pozitive Expiratory Pressure) — The device will be built according to the optimal design parameters for a positive expiratory pressure therapy bottle device established by Mestriner et al. According to this
  Bottle-P.E.P. device:
  * PEP: 10-20 cmH2O
  * Inspiration: Expiration Ratio: 1:3-4
  * Material Used: Open top plastic bottle, plastic pipe.
  Plastic Bottle Specifications:
  I. Material-Hard Plastic II. Dimensions-Weight- 40grams; Height- 25cm; Width- 10cm; Perimeter- 20cm III. Water column height- 13cm
  Plastic Pipe Properties:
  I. Material-Pipette II. Inner Diameter- ≥8mm III. Pipe Length- 30cm IV. Depth in the water column - 10cm; 3 cm above the bottom of the bottle surface.
  - The distal end of the tube used in the Bottle P.E.P. will be placed 10 cm below the surface, i.e. 10 cm water column and 3 cm above the bottom of the bottle, and the device will be placed on a table in front of the participant.
  Arms: Group II
Other: Early Mobilization — The Maebashi mobilization protocol will be followed for early mobilization program. According to this protocol, the hemodynamic and respiratory parameters of the patient will be evaluated first and the patient who meets the criteria for the mobilization program will be started to the mobilization program according to the appropriate stage of the 5-stage mobilization protocol.
  In Maebashi Mobilization protocol:
  Level 1: No mobilization and in-bed passive exercise Level 2: Supported in-bed sitting and in-bed active/assistive-active exercise Level 3: Unassisted sitting on the edge of the bed Level 4: Active transfer to chair Level 5: Standing, stepping in place and supported walking about 10 meters (with support of 2 people)
  Arms: Group III

SUMMARY:
The aim of this study was to investigate the effects of postoperative early mobilization and Bottle-P.E.P. application on respiratory parameters and functional capacity in patients undergoing heart valve surgery.

DETAILED DESCRIPTION:
After all patients were informed about the study and potential risks, patients who gave informed consent will be evaluated preoperatively and 5-7 days after surgery by the same investigator. Patients will be randomly divided into 3 groups: Group I (n=20, control) - conventional cardiopulmonary rehabilitation, Group II (n=20), conventional cardiopulmonary rehabilitation and Bottle P.E.P. application, Group III (n=20) will be included in the study as conventional cardiopulmonary rehabilitation and early mobilization group. The respiratory parameters of the patients will be determined by a pulmonary function test and their functional capacities will be determined by a 6-minute walk test. The preoperative and postoperative periods will be compared with statistical methods in the light of these evaluations on days 5-7.

ELIGIBILITY:
Inclusion Criteria:

* After heart valve surgery: Patients undergoing valvular surgery via sternotomy
* Same surgical technique (from med-sternum)
* Age group (25-75 Y)
* Stable hemodynamic values (stable vital signs, normal temperature, etc.)
* Full awareness of time and space

Exclusion Criteria:

* Ejection Fraction 35 %
* Any Male/female patient <25 or >75
* Body Mass Index (BMI) ≥ 38 kg/m2
* Intubation time >6 hours after surgery
* Uncontrolled arrhythmias
* Rheumatoid arthritis, other inflammatory and autoimmune diseases
* Active malignancy
* Cardiac pacemaker or defibrillator
* Mental health disorders
* Any postoperative complication (general muscle weakness, wound infection of the sternum or leg, stroke.)
* Refusal to assist in data collection

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-01-29 (Estimated); Study Completion 2025-01-29 (Estimated)

PRIMARY OUTCOMES:
European System for Cardiac Operative Risk Evaluation (EuroSCORE): | Preoperative period
  Mortality Risk Assessment is a risk scoring system used to predict mortality in the preoperative period in cardiac surgery.
  EuroSCORE: 0-3 points will be considered Low risk, 4-6 points will be considered Medium risk, 7 and above will be considered High risk.
New York Heart Association (NHYA) Functional Class Assessment: | Preoperative period
  The severity of symptoms in heart failure can be graded according to the amount of exertion that produces the symptom. It is a classification that grades heart failure into four separate classes in order to evaluate the effects of heart failure on functional capacity.
  NYHA Classification - The Stages of Heart Failure:
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Respiratory function test: | Preoperative 1st and 7th days
  Patients will be evaluated with spirometric measurements according to the American Thoracic Society and European Respiratory Society guidelines. Absolute values of FEV1, and forced vital capacity (FVC) were obtained, and their percent of the predicted values (% pred) were calculated .
  An obstructive spirometric pattern was defined as FEV1/FVC < 70%, and a restrictive spirometric pattern was defined as both FEV1/FVC ≥ 70% and FVC < 80% pred.
Baseline transthoracic echocardiography: | Preoperative 1st and 7th days
  Diastolic dysfunction and reduced ejection fraction (≤ 54% in females, and ≤ 52% in males) were defined according to the current guidelines.
  Interventricular septal thickness (IVSd), posterior wall thickness (PWd), and LV dimension (LVEDD) were all measured at end-diastole.
  The LV mass (LVM) was calculated according to the Deveraux formula using these measurements: LVM (g) = 0.80 × {1.04[(IVSd + LVEDD + PWd)3-(LVEDD)3]} + 0.6. LVM-index (LVMI) was calculated by dividing LVM by body surface area (BSA). BSA was calculated with the Mosteller formula.
  LV hypertrophy (LVH) was defined as LVMI ≥ 102 g/m2 for males and ≥ 88 g/m2 for females
NT-ProBNP measurement: | Preoperative 1st and 7th days
  NT-proBNP levels are useful in diagnosing heart failure and monitoring treatment effectiveness. High NT-proBNP levels may increase the severity or risk of heart failure.
  Normal values; For NT-proBNP, <125 pg/ml (<450 pg/ml over 75 years of age) is acceptable.
Functional capacity assessment: | Preoperative 1st and 7th days
  The 6 Minute Walk Test (6MWT) will be performed according to the recommendations of the American Thoracic Society. Patients will be instructed to walk the longest distance at the fastest speed possible for a period of 6 minutes. The length of the walking track will be 30 m. The physical therapist will provide standard stimulation every minute. If necessary, the patient will be allowed to rest during the test and this time will be included in the total test time. The test will be performed twice with 1-hour intervals between tests. The best distance will be recorded. The minimum clinically significant difference considered will be 25 m.
The Borg Category-Ratio scale (Borg CR-10) and The Modified Borg Dyspnea Scale (MBS): | Preoperative 1st and 7th days
  The Borg CR10 is a general intensity scale with specific bases for measuring effort and fatigue. Participants will be asked to mark their perceived level of fatigue on a vertical scale from 0 to 10 before and after the six-minute walk test.
  The Modified Borg Dyspnea Scale (MBS) is a 0 to 10 numerical score used to measure self-reported dyspnea during submaximal exercise. Participants will be asked to circle or mark the number that best describes their level of dyspnea before and after the six-minute walk test.
Functional Independence Measurement (FIM): | Preoperative 1st and 7th days]
  The level of independence in daily living activities is an assessment tool used to evaluate the patient's functional status throughout the rehabilitation process.
  FIM is divided into two domains: Motor and Cognitive. It consists of a total of 18 items, 13 items in the motor domain and 5 items in the cognitive domain. Each item in the FIM is scored on a 7-point Likert scale, and the score indicates the amount of assistance required to accomplish each item. 1 = activities are done completely dependently, 7 = activities are done independently by the individual. A final total score is created and individuals' scores range from 18-126, where a score of 18 represents the individual is completely dependent and 126 represents complete independence.
Visual Analog Scale - Pain Assessment: | Preoperative 1st and 7th days
  Visual Analog Scale (VAS) was used to assess the pain severity of the patients. Chest pain before the operation and incision site pain in addition to chest pain after the operation will be questioned.
  The minimum clinical significance level for the scale (Minimal clinically important differences) will be taken as an MCID value of 3. VAS is a subjective pain assessment scale that determines pain levels by having patients mark the point where they feel their pain on a 10-centimeter horizontal line.
  Marked on the scale are 0 - no pain, 10 - unbearable pain. The marked point will be measured with a ruler and recorded.

SECONDARY OUTCOMES:
RASS (Richmond Agitation and Sedation Scale): | Postoperative 1st day in intensive care unit
  It will be used for Agitation, Anxiety and Sedation Assessment. RASS score is a 10-point scale with points between +4 and -5. +1 and +4 points indicate the presence and severity of anxiety and agitation, 0 points indicate alertness and calm, -1 and -5 points indicate sedation level. If RASS is ≤ -3 or >+2: A consultation will be held with the specialist physician about starting rehabilitation, and after the patient's sedation and analgesic medical treatment is arranged, the decision to start rehabilitation will be made with the approval of the patient-physician.
  RASS ≤ -2 or <+1 rehabilitation will begin. An evaluation will be performed before treatment in the intensive care unit on the first postoperative day.
Evaluation of hemodynamic and respiratory parameters: | Postoperative 1st day
  1. Heart Rate
     * Unit of Measure: Beats per minute (bpm)
     * Normal Range: 60-120 bpm
  2. Systolic Blood Pressure
     * Unit of Measure: Millimeters of mercury (mmHg)
     * Normal Range: >90 and <200 mmHg
  3. Respiratory Rate
     * Unit of Measure: Breaths per minute (b/min)
     * Normal Range: <35 b/min
  4. Inspired Fractional Oxygen Amount (FiO2)
     * Unit of Measure: Percentage (%)
     * Calculation: FiO2 (%) = 21 + (L/min Oxygen x 4)
     * Normal Range: ≤60%
  5. Positive End-Expiratory Pressure (PEEP)
     * Unit of Measure: Centimeters of water (cmH2O)
     * Normal Range: ≤10 cmH2O
  6. Oxygenation Adequacy
     * Unit of Measure: Percentage (%)
     * Normal Range: SaO2 ≥90%
  7. Gas Exchange and Oxygenation Status (PaO2/FiO2 Ratio)
     * Unit of Measure: Millimeters of mercury (mmHg)
     * Normal Range: 300-500 mmHg
     * Abnormal Range: <300 mmHg indicates abnormal gas exchange, <200 mmHg indicates severe hypoxemia
  8. Vasopressor Use • Unit of Measure: Dosage amount
Arterial blood gas measurements: | Postoperative 1st day in intensive care unit
  Oxygenation will be calculated by recording the PaO2/FiO2 ratio from arterial blood gas samples taken in the intensive care unit on postoperative day 1, before the mobilization program and 30 minutes after recovery.
  Normal PaO2/FiO2 ratio of 300-500 mmHg is considered normal. Values <1300 mmHg indicate abnormal gas exchange, and <200 mmHg indicate severe hypoxemia.
  FiO2 (%)= 21 + (L/min Oxygen x 4)
Postoperative complication evaluation: | Postoperative 1st and 7th days
  It will be diagnosed by the clinician if one or more of the following criteria are present:
  1. pneumonia-presence of radiological evidence of pulmonary infiltration associated with at least two findings including purulent sputum, elevated body temperature (>38.0°C) or leukocytosis (⩾25% above preoperative baseline);
  2. tracheobronchitis-marked increase in sputum production or presence of purulent sputum in a patient with a normal chest X-ray;
  3. atelectasis with clinical implications-radiological evidence of lung atelectasis associated with dyspnea;
  4. Hypoxemia and oxygen demand below SpO2 < 85%;
  5. Acute respiratory failure-acute lack of gas exchange requiring invasive or noninvasive mechanical ventilation.
  6. Permanent stroke
  7. Postcardial tamponade
  8. Postoperative delirium
Length of hospital stay: | Duration of hospital stay
  Hospital stay (evaluated up to 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Rezan Aksoy, Ass Prof Dr, Study Chair — Istanbul Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital; Recep Çalışkan, Doctor, Study Chair — Istanbul Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Locations (1):
- Istanbul Provincial Health Directorate Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Education Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No